CLINICAL TRIAL: NCT04300686
Title: A Pilot Study in the Treatment of Severe Patients With Takayasu Arteritis With Tocilizumab and Adalimumab, Based on ECTA Cohort
Brief Title: A Pilot Study in Severe Patients With Takayasu Arteritis.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TACTIC-SS
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Takayasu Arteritis; Tocilizumab; Adalimumab; Treatment
Keywords: Takayasu Arteritis; Tocilizumab; Adalimumab; treatment
MeSH Terms: conditions — Takayasu Arteritis | interventions — tocilizumab; Adalimumab

STUDY DESIGN:
Intervention Model Description: Severe TAK patients were divided into two groups, with 20 cases for each group at the randomized ratio 1:1, prescribed with adalimumab (40mg.bim.IH) and tocilizumab (8mg/kg.qm.ivgtt) respectively, in the presence of prednisone. After the 24 weeks of treatment, the disease remission is evaluated (primary endpoint). If the disease activity is alleviated (remission), the strategy would be maintained for another 24weeks, otherwise (resistant), the treatment strategy would be shifted to the opposite for 24weeks. After 48 weeks, the disease remission would be evaluated once again (secondary endpoint).
Masking Description: None. Open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tocilizumab (Active Comparator): This group of 20 TAK cases are prescribed with tocilizumab (Dose: 8mg/kg. qm. ivgtt.) for 24 weeks.
  Interventions: Biological: Tocilizumab
- Adalimumab (Experimental): This group of 20 TAK cases are prescribed with adalimumab (Dose: 40mg.bim.IH.) for 24 weeks.
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Tocilizumab — The tocilizumab group is prescribed with tocilizumab (8mg/kg.qm.ivgtt.) for 24 weeks, and the disease activity is monitored in the follow-up (primary endpoint).
  After 24 weeks of treatment, if the disease is alleviated (remission), then the usage of tocilizumab is maintained for another 24 weeks, otherwise (resistant), patients would be given adalimumab (40mg.bim.IH.) for 24 weeks instead.
  Other Names: IL-6R alpha antibody
  Arms: Tocilizumab
Biological: Adalimumab — The adalimumab group is prescribed with adalimumab (40mg.bim.IH) for 24 weeks, and the disease activity is monitored in the follow-up (primary endpoint).
  After 24 weeks of treatment, if the disease is alleviated (remission), then the usage of adalimumab would be maintained for another 24 weeks, otherwise (resistant), patients would be given tocilizumab (8mg/kg.qm.ivgtt.) for 24 weeks instead.
  Other Names: TNF-alpha antibody
  Arms: Adalimumab

SUMMARY:
Takayasu arteritis (TAK) is a rare chronic inflammatory arteritis, which lacks an effective well-accepted intervention strategy. We classify TAK patients into 3 levels, including mild, moderate, and severe. And the biological agents tocilizumab and adalimumab are randomly prescribed in severe patients, to find out the relatively better treatment strategy, facilitating better intervention strategy in severe TAK patients.

DETAILED DESCRIPTION:
The Takayasu arteritis (TAK) is a rare chronic inflammatory arteritis, which lacks an effective well-accepted intervention strategy. Previous studies have revealed that methotrexate, tofacitinib, adalimumab, and tocilizumab were effective in controlling disease activity and preventing disease relapse in some TAK patients, especially the latter two biological agents. However, we believed that different patients should be prescribed different drug combinations, i.e. personalized medicine, to obtain the optimal intervention effect.

Here we tried to classify the TAK patients into three levels including mild, moderate, and severe, and prescribe different drug interventions to discover which biological agent is better in severe TAK patients.

1. Patients were classified as mild, moderate, and severe groups according to the disease severity of TAK patients.

1.1 Severe

1. Severe hypertension

   1. Continuously upper limb systolic blood pressure ≥180mmHg or diastolic blood pressure ≥110mmHg;
   2. OR upper limb blood pressure cannot be measured if lower limb systolic blood pressure ≥200mmHg or diastolic blood pressure ≥120mmHg;
   3. With target organ damage due to hypertension;
2. Aortic arch and its branches involved

   a. Multiple branches involved (two or more) and severe stenosis (stenosis rate ≥70%); b. stenosis rate ≥50%, accompanied by nervous system ischemic symptoms and/or signs; c. stenosis rate ≥50%, accompanied by a recent history of cerebrovascular events;
3. The carotid artery and its branches involved

   1. Multiple branches (two or more) involved and severe stenosis (stenosis rate ≥70%);
   2. stenosis rate ≥50%, accompanied by nervous system ischemic symptoms and/or signs;
   3. stenosis rate ≥50%, accompanied by the recent history of cerebrovascular events;
4. Pulmonary artery involvement

   a. Chest tightness, hemoptysis, dyspnea, radionuclide pulmonary ventilation/blood perfusion imaging or CTA suggesting pulmonary artery thrombosis with respiratory failure (type I); b. Chest tightness, shortness of breath, and cardiac ultrasound suggesting severe pulmonary artery hypertension with cardiac function abnormality (NYHA class III and above);
5. The coronary artery involved

   1. The onset of unstable angina pectoris or myocardial infarction;
   2. Cardiac ultrasound indicating ischemic cardiomyopathy, NYHA class III and above;
6. The aortic valve and aortic root involved

   1. Severe reflux of the aortic valve;
   2. OR aortic valve leakage, annulus tearing;
   3. OR aneurysm in the aortic root and/or ascending aortic (≥2 times in diameter);
   4. OR dilation of the aortic root and/or ascending aorta (≥5cm in diameter);
   5. OR dissection of the aortic root and/or ascending aorta; Any item of the above a - e is accompanied by abnormal cardiac function (NYHA III and above);
7. Renal artery involved a. Severe stenosis of renal artery secondary to malignant hypertension (blood pressure is still 180 / 120mmHg after treatment with three or more antihypertensive drugs) b. Severe renal artery stenosis accompanied by a progressive increase in serum creatinine or a reduction in glomerular filtration rate (GFR) of ≥25%;
8. Glucocorticoids and the traditional synthetic chemical immunosuppressants were of no use. And the disease is not well controlled with the severe injury of the organs.

1.2 Moderate

1. Hypertension

   a. Upper limb systolic blood pressure ≥160-180mmHg or / and diastolic blood pressure ≥100-110mmHg; b. OR upper limb blood pressure is unmeasurable or lower limb systolic blood pressure is ≥180mmHg or diastolic blood pressure is ≥100-110mmHg;
2. Aortic arch and its branches involved

   a. 1-2 vessels are involved with moderate stenosis (stenosis rate ≥50%-<70%); b. Dizziness occurs during physical activity, and symptoms disappear in the resting state;
3. The carotid artery and its branches involved

   a. Unilateral or bilateral vascular stenosis rate ≥50% -70%, with dizziness during light physical activity;
4. Pulmonary artery involved

   a. Radionuclide pulmonary ventilation/blood perfusion imaging or CTA indicates pulmonary vascular disease; chest tightness after activity; Cardiac ultrasound indicates moderate pulmonary artery hypertension (pressure> 40-60mmHg), with abnormal cardiac function (NYHA class Ⅱ);
5. Coronary artery involvement

   a. Chest tightness and chest pain after moderate activities, CTA showed 50% or more in coronary artery stenosis, abnormal cardiac function (NYHA class Ⅱ);
6. The aortic valve and aortic root involved

   1. Moderate aortic regurgitation;
   2. Aortic root and/or ascending aortic aneurysm (diameter <2 times);
   3. Dilation of the aortic root and/or ascending aorta (diameter <5cm); Each item of a - c is accompanied by abnormal cardiac function (NYHA Class II);
7. Renal artery involvement a. Renal artery stenosis rate ≥50%, and blood pressure 160-180 / 110-120 (excluding 120) mmHg after treatment, or with left ventricular myocardial hypertrophy, hypertension and heart disease, CKD-II;

1.3 Mild

1. Hypertension

   1. Upper limb systolic blood pressure ≥140mmHg or diastolic blood pressure ≥90mmHg;
   2. OR upper limb blood pressure is unmeasurable or lower limb systolic blood pressure is ≥140mmHg or diastolic blood pressure is ≥90mmHg;
2. Aortic arch and its branches involved a. Single or multiple lesions with mild stenosis (stenosis rate <50%), and without neurological ischemic symptoms and/or signs in daily activities;
3. The carotid artery and its branches involved

   a. Single or multiple lesions with mild stenosis (stenosis rate <50%) and no neurological ischemic symptoms and/or signs during daily activities;
4. The pulmonary artery involved

   1. Cardiac ultrasound indicates mild or normal pulmonary artery pressure (pressure 30-40mmHg);
   2. Imaging shows pulmonary arteritis or pulmonary artery stenosis, occlusion a and b, with chest tightness, shortness of breath, and hemoptysis without activity; cardiac function (NYHA I), normal blood gas analysis;
5. The coronary artery involved

   a. Chest tightness, shortness of breath, chest pain after inactivity; cardiac function (NYHA I);
6. The aortic valve and aortic root involved

   1. Mild aortic regurgitation;
   2. Aortic root and / or ascending aortic aneurysm-like expansion (diameter <1.5 times); a and b, each with cardiac function (NYHA I);
7. Renal artery involved a. Renal artery stenosis rate <50%, without/with mild hypertension (see 1), or normal serum creatinine, normal or slightly impaired glomerular filtration rate (GFR);

1.2. Based on the TAK patients in the ECTA cohort (Clinical trials. No: NCT03893136), we tried to compare the treatment efficacy of biological agents between tocilizumab (TCZ) and adalimumab (ADA) in severe TAK patients, with a pilot study.

Other important detailed description of the study are listed as follows:

1. Basic treatment of prednisone:

   The initial prednisone dose is 40mg.qd.po, and maintained for 1 month. After 1 month's treatment, the dose is gradually tapered to 15mg by 5mg per 2 weeks. Subsequently, the dose is decreased to 5mg by 2.5mg per 3 months. The 5mg is the final target maintained dose. In the treatment, if the relapse occurs, the dose of prednisone returned to the last dosage. For example, if the patient gets a relapse at the dose of 15mg of prednisone, then the dose of prednisone returned to 20mg.

   The relapse of TAK is defined according to the "2018 Update of the EULAR recommendations for the management of large vessel vasculitis". Relapse includes major relapse or minor relapse. Major relapse: Recurrence of active disease with either of the following: a. Clinical features of ischemia* (including jaw claudication, visual symptoms, the visual loss attributable to TAK, scalp necrosis, stroke, limb claudication). b. Evidence of active aortic inflammation resulting in progressive aortic or large vessel dilatation, stenosis or dissection. Minor relapse Recurrence of active disease, not fulfilling the criteria for the major relapse.
2. ADA: 40mg bim IH.
3. TCZ: 8mg/kg qm ivgtt.
4. Treatment shift: if the TAK patients in ADA group failed to reach clinical remission at the end of 24th week, they would be shifted to TCZ group starting a new round of induction and complete the rest 24-week follow-up; and vice versa;

In the follow-up, the disease remission and related markers are monitored.

ELIGIBILITY:
Inclusion Criteria:

1. age≥14 years old;
2. active: Kerr score≥ 2;
3. severe:

   1. Blood pressure > 180/110mmHg;
   2. ≥ 3 branches with the stenotic rate > 70% involved;
   3. high degree of organ insufficiency: NYHF III~IV; eGFR (MRDR) 15~ 60ml/min;

Exclusion Criteria:

1. Severe organ insufficiency;
2. Acute or chronic active infections including tuberculosis, hepatitis virus, etc.;
3. Other autoimmune diseases including systemic lupus erythematosus, Behcet disease, IgG4 relative disease;
4. malignant tumors;
5. history of severe drug allergy;
6. successive twice relapse occurs even after the intervention adjustment ( for the benefits of patients)

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease remission at 24 weeks. | 24 weeks
  comparison of clinical remission rate between adalimumab and tocilizumab groups at the end of 24th week follow-up;

SECONDARY OUTCOMES:
Disease remission at 48 weeks. | 48 weeks
  comparison of clinical remission rate between adalimumab and tocilizumab groups at the end of 48th week follow-up;
Prednisone dose reduction at endpoint | 24 weeks and 48 weeks.
  comparison of targeted prednisone usage between adalimumab and tocilizumab groups at the end of 24th and 48th week follow-up;
disease relapse in the follow-up | At the time point of 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks, 36 weeks, 48 weeks.
  comparison of disease relapse between adalimumab and tocilizumab groups; (Relapse is defined as: (1) Major relapse: Major relapse Recurrence of active disease with either of the following: a. Clinical features of ischaemia* (including jaw claudication,visual symptoms, visual loss attributable to TAK, scalp necrosis, stroke, limb claudication). b. Evidence of active aortic inflammation resulting in progressive aortic or large vessel dilatation, stenosis or dissection. (2) Minor relapse: Recurrence of active disease, not fulfilling the criteria for a major relapse.)
Vascular progression in angiographic examination at 6 months and 12 months. | 24 weeks and 48 weeks.
  comparison of vascular change with MRA, CTA, or doppler ultrasound angiographic examinations between adalimumab and tocilizumab groups;
Change of the quality of life with questionnaire SF-36 | At the time point of 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks, 36 weeks, 48 weeks.
  comparison of quality of life between adalimumab and tocilizumab groups with the 36-Item Short Form Health Survey questionnaire (SF-36) (Scores:0~100, lower score means more disability)
Change of the quality of life with questionnaire MOS-sleep scale | At the time point of 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks, 36 weeks, 48 weeks.
  comparison of quality of life between adalimumab and tocilizumab groups with the questionnaire of sleep scale from medical outcomes study (MOS-sleep scale) (Scores: 11-65, lower scores indicates more difficulty in sleep)
Change of the quality of life with the Fatigue severity scale | At the time point of 2 weeks, 4 weeks, 8 weeks, 12 weeks, 16 weeks, 20 weeks, 24 weeks, 36 weeks, 48 weeks.
  comparison of quality of life between adalimumab and tocilizumab groups with the Fatigue severity scale (Scores: 9-63, higher score means severe fatigue)

CONTACTS AND LOCATIONS:
Overall Officials: Lindi Jiang, PhD, Study Chair — Fudan University
Locations (1):
- Department of Rheumatology in Zhongshan hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Kong X, Ma L, Ding Z, Chen H, Chen R, Jin X, Chen C, Lin J, Jiang L. Treatment efficacy and safety of adalimumab versus tocilizumab in patients with active and severe Takayasu arteritis: an open-label study. Rheumatology (Oxford). 2024 May 2;63(5):1359-1367. doi: 10.1093/rheumatology/kead387. PMID 37540159

DOCUMENTS (1):
  • Study Protocol (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT04300686/Prot_000.pdf